CLINICAL TRIAL: NCT05664425
Title: Mechanical Treatment of Peri-Implant Mucositis -the Effect of Submucosal Instrumentation
Brief Title: Mechanical Treatment Peri-Implant Mucositis
Acronym: MechTreatPiM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Anders Verket, Principal investigator, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MechTreatPiM
Record Dates: First submitted 2022-12-08; First posted 2022-12-23 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Peri-implant Mucositis

STUDY DESIGN:
Intervention Model Description: Parallell group two-arm randomised study
Who Masked: Investigator
Masking Description: Investigator-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanical treatment arm + oral hygiene reinforcement (Experimental): Subjects receive oral hygiene reinforcement, and additionally submucosal instrumentation with ultrasonics with a plastic tip.
  Interventions: Device: Ultrasonic debridement
- Oral hygiene reinforcement alone (No Intervention): Subjects receive oral hygiene reinforcement, but do not receive submucosal instrumentation.

INTERVENTIONS:
Device: Ultrasonic debridement — Ultrasonic debridement with a plastic/teflon tip (2 minutes + 1 minute irrigation)
  Arms: Mechanical treatment arm + oral hygiene reinforcement

SUMMARY:
This two-arm, single-blinded, monocentric, controlled, randomised clinical study is designed to examine the effect of professional submucosal treatment by means of ultrasonics with plastic tip (test group), as compared to no professional submucosal instrumentation (control group), in the treatment of peri-implant mucositis (PIM). Both groups will have oral hygiene instruction/reinforcement (OHI) at baseline and repeated at 3 months. In the study, 50 participants will be enrolled (25 per group), with each patient contributing one implant with PIM. Peri-implant sulcus fluid (PISF) samples will be obtained at baseline, 3- and 6-months to analyse the change of relevant biomarkers over the course of PIM treatment. Intraoral scans will be performed at baseline, 3- and 6-months to analyse potential soft-tissue volumetric changes according to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥ 20 years
* Subject must have one implant presenting PIM as defined according to the World Workshop 2017 criteria (presence of BoP and/or suppuration (SoP), without bone loss exceeding 0.5 mm beyond crestal bone level changes resulting from initial remodeling, regardless of PPD. In absence of baseline radiographs (i.e., 0-1 year after loading) a bone level of <2mm from the top of the intraosseous part of the implant is considered as the reference threshold)
* Cleansable prosthesis (an interproximal brush must be able to pass from side to side at interproximal aspects tangential to the peri-implant sulcus, and a brush has to be able to reach the buccal and palatal/lingual sulcus).
* No evidence of occlusal overload
* No cement remnants identified on radiographs or clinically
* Implant-supported fixed restoration inserted at least 6 months before patient enrolment and not interfering with assessment of clinical parameters at more than 3/6 sites
* Periodontally healthy subjects or treated periodontitis (no residual site with PPD ≥ 5 mm)
* Full-mouth plaque (FMPS) and bleeding (FMBS) score ≤ 20%¬¬¬¬¬¬¬ at screening visit
* Non-smokers or light-smokers (<10 cigarettes per day)
* Competent to give consent

Exclusion Criteria:

* Previous radiotherapy, current use of chemotherapy, systemic long-term corticosteroid treatment
* Hematologic disorders
* Pregnant subjects
* Patients classified as > class 2 according to the ASA (American Society of Anesthesiologists) physical status classification
* No systemic antibiotic treatment within 3 months prior to intervention

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Bleeding on probing (BoP) extent | 6 months
  Reduction in the extent of BoP as measured on six sites per implant

SECONDARY OUTCOMES:
Peri-implant sulcus fluid (PISF) biomarkers | 6 months
  Biomarkers sampled at baseline, 3- and 6-months
Intraoral digital scan | 6 months
  Volumetric change of soft tissue following peri-implant mucositis treatment
Disease resolution | 6 months
  No BoP at any of the six probed sites at 6-month follow-up
Severity of BoP | 6 months
  Reduction in the severity of BoP (graded from 0-3) at 6 months
Probing pocket depth (PPD) reduction | 6 months
  Reduction in PPD at 6 months
Bone level changes | 6 months
  Changes in bone level as assessed by radiographs at baseline and 6-months
Onset of peri-implantitis | 6 months
  If peri-implantitis is diagnosed during or following the study, this will be reported. Peri-implantitis is defined as progressive bone loss identified by an increase of PPD changes or bone level changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Clinical Dentistry, Faculty of Dentistry, University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
IPD will be available for other researchers upon reasonable request and as long as in accordance with ethical committee and national GDPR rules.